CLINICAL TRIAL: NCT01025401
Title: Caractérisation et détection Des Mouvements Durant Les Crises d'épilepsie à Des Fins d'Alarme, Pour un Usage en Institution et en Famille.
Brief Title: Characterization of Epileptic Motor Patterns by Tridimensional Analysis of Movement 2
Acronym: CAPAMETRIM2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: departure of a collaborator in charge of the data collection
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Philippe KAHANE/MD-PHD, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0905; 2009-A00196-51 (Registry Identifier: ID RCB)
Record Dates: First submitted 2009-06-29; First posted 2009-12-03 (Estimated); Last update posted 2010-11-23 (Estimated); Status verified 2010-11

CONDITIONS: Epileptic Patients With Motor Manifestations During Seizures
Keywords: epilepsy; seizures; movement
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motor manifestations during seizures (No Intervention)
  Interventions: Device: 3-D accelerometric and magnetic sensors

INTERVENTIONS:
Device: 3-D accelerometric and magnetic sensors — sensors are positioned on the right wrist, the left wrist and on the head.

SUMMARY:
CAPAMETRIM 2 aims to characterize epileptic motor patterns by a quantitative three-dimensional analysis of movements.

This is done to obtain a 3-D motor signature of seizures, for a given patient, and allows their detection with an ambulatory monitoring system.

The benefit for patients is to improve the diagnosis of their diseases by better characterizing their seizures.

DETAILED DESCRIPTION:
CAPAMETRIM 2 aims to characterize epileptic motor patterns by a quantitative three-dimensional analysis of movements.

The project is planned in three phases:

* Installation of 3-D accelerometric and magnetic sensors acquisition systems on the hospital (extension of a preceding study CAPAMETRIM).
* Collection of data on epileptic patients. Sensors will be positioned on the right and left hands and on the head. A 3-D analysis of movements will be done according to the collection by tagging data with visual analysis made on video.
* Development of a motor pattern classification system used for seizure detection.

ELIGIBILITY:
Inclusion Criteria:

* Adult or children (>= 6 years)
* Written inform consented from the patient or its legal representative
* Presurgical investigation of pharmaco-resistant partial epilepsy
* Motor manifestations during seizures

Exclusion Criteria:

* Proved generalized epilepsy
* No motor manifestations during seizures
* Pregnant women
* Subjects deprived of freedom by an administrative or judicial decision

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
3-D accelerometric and magnetic sensors | continuously during hospitalization recordings (46 Hz from 9 h to 17 h)

SECONDARY OUTCOMES:
Video | continuously during hospitalization recordings (25 fps from 9 h to 17 h)
EEG | continuously during hospitalization recordings (256-1024 Hz from 9 h to 17 h)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Kahane, MD PHD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Grenoble University Hospital Epilepsy Monitoring Unit, Grenoble, France